CLINICAL TRIAL: NCT02593734
Title: Joining Forces: Integrating Psychotropic Medication Into the Care of People With Mental Disorders in a Prayer Camp in Ghana
Brief Title: Integrating Psychotropic Medication Into the Care of People With Mental Disorders in a Prayer Camp in Ghana
Acronym: JFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ghana Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JFR
Record Dates: First submitted 2013-11-25; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia; Mood Disorders,; Anxiety Disorder
MeSH Terms: conditions — Schizophrenia; Mood Disorders; Anxiety Disorders | interventions — Olanzapine; Risperidone; Amitriptyline; Fluoxetine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No intervention
- Experimental (Experimental): The intervention is prescription and dispensing by a nurse of oral antipsychotic or antidepressant medication as clinically indicated. The mediations to be selected from include oral olanzapine, risperidone, amitryptaline or fluoxetine at doses prescribed by the treating psychiatrist.
  Interventions: Drug: olanzapine; Drug: risperidone; Drug: amitryptaline; Drug: fluoxetine

INTERVENTIONS:
Drug: olanzapine — oral antipsychotic drug therapy
  Other Names: Zyprexa
  Arms: Experimental
Drug: risperidone — oral antipsychotic drug therapy
  Other Names: Risperdal
  Arms: Experimental
Drug: amitryptaline — oral antidepressant drug therapy
  Other Names: Elavil
  Arms: Experimental
Drug: fluoxetine — oral drug therapy for depression
  Other Names: Prozac
  Arms: Experimental

SUMMARY:
The purpose of this study is to evaluate a bundled intervention of psychotropic drugs and daily contact with a nurse for people with mental health disorders in a prayer camp and secondly to assess whether the attitudes of the prayer camp staff toward mental health disorders and conventional medicines remain the same after the intervention.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a bundled intervention of psychotropic drugs and daily contact with a nurse for people with mental health disorders in a prayer camp and secondly to assess whether the attitudes of the prayer camp staff toward mental health disorders and conventional medicines remain the same after the intervention.

In the proposed study, residents of the sanatorium at the Mount Horeb Prayer Center located in Mamfe, Ghana will be screened for psychiatric disorders by a psychiatrist. Those who are diagnosed with a psychiatric disorder requiring treatment (schizophrenia, or mood disorder) and who meet the other inclusion criteria (see below) will be randomly assigned to receive a daily dose of the appropriate psychotropic drug (according to standard procedures of care) as well as regular prayer camp treatment (intervention group) or to receive only regular prayer camp treatment (control group). After randomization, the patients in the intervention group will receive the bundled treatment for 6 weeks, while control group patients will receive regular prayer camp treatment, e.g. encouragement to pray. Psychiatrists blinded to group assignments will assess outcomes over a 6 - 8 week period. Following this, patients will be referred for continued care with health care facilities as close to their homes as possible on discharge and if they so desire. At the start of the intervention, pastors and attendants at the prayer camp will be qualitatively assessed through a semi-structured interview concerning their attributions of mental illness causation. They will be assessed -0, -6 weeks after and again -12 weeks after intervention. The investigators hypothesize that patients who receive the bundled intervention will have improved mental health outcomes and functioning and that prayer camp staff will develop more positive attitudes toward conventional medicine and will begin to conceptualize mental health disorders as treatable illnesses, rather than only as a spiritual disorder. The results will provide empirical evidence for or against an integrated model of community based care which encompasses the medical and spiritual. This is the first intervention study in Sub-Saharan Africa to promote the use of psychotropic drugs in a traditional or spiritual healing setting. Its findings may inform the implementation of national policies governing collaboration between primary health care and faith healing centers, expanding access to and improving the quality of mental health care services.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years,<70
2. Will benefit from treatment
3. Not suffering from physical condition
4. Resident at the prayer camp
5. Not likely to be discharged from camp within six weeks
6. Speaks either English or twi
7. Able to give consent
8. Not already on medication

Exclusion Criteria:

1. likely to be discharged within 6 weeks of commencement of medication
2. Patients already on medication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Brief Psychiatric Rating Scale (BPRS) | 6 weeks

SECONDARY OUTCOMES:
Clinical Global Impressions(CGI) | 6 weeks
Global Assessment of functioning(GAF) | 6 weeks
De-chaining, | 6 weeks
  The number of days in each week that the patient was NOT restrained with physical restraints such as chains

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Ofori-Atta, PhD, Principal Investigator — University of Ghana Medical School
Locations (1):
- Mount Horeb Prayer Centre, Mamfe, Ghana

REFERENCES:
- [Derived] Ofori-Atta A, Attafuah J, Jack H, Baning F, Rosenheck R; Joining Forces Research Consortium. Joining psychiatric care and faith healing in a prayer camp in Ghana: randomised trial. Br J Psychiatry. 2018 Jan;212(1):34-41. doi: 10.1192/bjp.2017.12. PMID 29433613